CLINICAL TRIAL: NCT07051473
Title: Impact of Coronary CT Angiography Findings on Prognosis of Patients Undergoing Percutaneous Coronary Intervention
Brief Title: Relationship Between Coronary CT Angiography Findings and Prognosis Of Patients Undergoing PCI
Status: Recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Alpin Mert TEKİN, Research Assistant, Istanbul University - Cerrahpasa
Other Study IDs: 2025/66
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Vulnerable plaque; Vulnerable patient; Vulnerable blood; High risk coronary plaques; PCI; Coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High risk plaque features positive, PCI positive: The people that has at least one lesion in their coronary arteries, carrying at least one high-risk plaque feature, derived from CCTA and treated with PCI of that lesion
- High risk plaque features positive, PCI negative: The people that has at least one lesion in their coronary arteries, carrying at least one high-risk plaque feature, derived from CCTA and not treated with PCI of that lesion
- High-risk plaque features negative, PCI positive: The people that has no lesion in their coronary arteries, carrying at least one high-risk plaque feature, derived from CCTA and treated with PCI of any lesion

SUMMARY:
Researchers at Cerrahpaşa Medical School in Istanbul are studying how a heart imaging test called coronary CT angiography can help improve care for people with coronary artery disease. This disease happens when fatty buildups, known as plaques, form in the arteries that supply blood to the heart. Over time, these plaques can limit blood flow and lead to serious problems like heart attacks. The goal of this research is to better understand which types of plaques may lead to worse outcomes, and how treatment choices-such as placing a stent or using medication-can affect a person's long-term heart health. This study will help doctors make better treatment decisions in the future. Some plaques are more dangerous than others, even when they don't cause major blockages. These are called high-risk or "vulnerable" plaques. Even though they may not narrow the artery much at first, they can still cause heart attacks in the future. Currently, doctors do not usually place stents in arteries unless the plaque causes a serious blockage. This is because stenting also carries risks, and it is not clear whether treating high-risk plaques early-before they cause problems-helps people live longer or feel better. This study hopes to find out whether certain types of plaques should be treated differently in the future. This study will include at least 789 adults who have already had coronary CT angiography as part of their regular care at Cerrahpaşa Medical School's cardiology clinic. These participants were treated either with a stent or with medication, depending on their medical needs. The decision to do the scan and how to treat the person was made by their doctor, following national and international medical guidelines. People who join the study do so voluntarily. They can choose to leave the study at any time without affecting their regular medical care. Participants will be followed for at least one year, starting from the day of their CT scan. They will return for check-ups at 3, 6, and 12 months. After the first year, they will continue to have yearly follow-up visits as part of routine care. At each visit, the study team will check symptoms, such as chest pain or shortness of breath; monitor health indicators, like cholesterol and blood sugar; and review any new heart procedures or treatments. Researchers will also review results from medical tests, such as blood tests, electrocardiograms (EKGs), heart ultrasounds (echocardiograms), repeat heart scans or procedures if done. If a participant has had a heart procedure done at another hospital, they will be asked to bring those records to their next appointment. This helps the research team get a full picture of each participant's heart health. The researchers will look at the features of the plaques seen in each participant's heart scan. They want to find out which types of plaques are more likely to lead to heart attacks or other serious problems. Participants will be divided into groups based on whether they received a stent or not. The researchers will compare outcomes between these groups to see if certain plaque types are more dangerous and whether stenting made a difference. The study will try to answer questions like: which plaque features are linked to future heart problems; do people with high-risk plaques do better with stents or with medication; can doctors use plaque features to decide who should get a stent? This research may help doctors better identify high-risk plaques and choose the right treatment for each person. The study does not involve any new, experimental, or unapproved treatments. All participants will receive medical care that follows well-established guidelines from groups like the European Society of Cardiology (ESC) and the American Heart Association (AHA). Participants are not asked to take new medications or undergo any tests or treatments that are not already part of their usual care. If new medical knowledge becomes available during the study that could affect treatment, participants will be informed and can choose whether to continue with the original plan or make changes. All personal and medical information will be kept confidential. The data will be stored securely in the hospital's system, and only the research team and authorised health officials will be allowed to access it. Participants' names and other identifying information will not appear in any published reports. If a participant wants to know their results or the overall results of the study, they can ask for a report. Even if someone leaves the study or stops coming to the clinic, the information already collected may still be used in the research unless the participant requests otherwise. There is no cost to participate in this study. The study will not affect your health insurance or create any additional charges. All medical care will continue to be covered by Turkey's national health system or your existing insurance.

ELIGIBILITY:
Inclusion Criteria:

1. Be over 18 years of age.
2. Have presented to the Cardiology Department of Cerrahpaşa Medical Faculty with symptoms or findings suggestive of stable coronary artery disease and undergone a coronary CT angiography based on clinical evaluation.
3. In addition, meet at least one of the following conditions:

   * The coronary CT angiography showed at least one lesion with at least one high-risk plaque feature, and based on the 2018 European Society of Cardiology (ESC) Guidelines on Myocardial Revascularisation and the presence of CAD-RADS 1 or 2 lesions, no revascularisation was performed.
   * The coronary CT angiography revealed a CAD-RADS 3 or higher lesion without high-risk plaque features, and revascularisation was performed on the target lesion, in accordance with the 2018 European Society of Cardiology (ESC) Guidelines on Myocardial Revascularisation.
   * The coronary CT angiography revealed a CAD-RADS 3 or higher lesion with high-risk plaque features, and revascularisation was performed on the target lesion, in accordance with the 2018 European Society of Cardiology (ESC) Guidelines on Myocardial Revascularisation.

Exclusion Criteria:

* Being underaged (below 18 years of age).
* Loss of medical follow-up data caused by discontinuation of participation in follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of individuals residing in the Republic of Turkey. The study sample was selected using a simple random sampling method and includes individuals from this population who presented to the Cardiology Department of Cerrahpaşa Medical Faculty with symptoms or findings suggestive of stable coronary artery disease. It is assumed that every citizen living within the borders of the Republic of Turkey has an equal probability of presenting to the clinic with complaints related to this condition.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
All cause death | Baseline, 3 months, 6 months, 12 months
  Death from any cause
Major adverse cardiovascular events | Baseline, 3 months, 6 months, 12 months
  Composition of cardiac death, spontaneous myocardial infarction, target vessel myocardial infarction, target vessel revascularisation, target lesion revascularisation

SECONDARY OUTCOMES:
Any myocardial infarction | Baseline, 3 months, 6 months, 12 months
  Any event of myocardial infarction defined by the "Fourth Universal Definition Of Myocardial Infarction"
Any revascularisation procedure | Baseline, 3 months, 6 months, 12 months
  Revascularisation by either percutaneous coronary intervention or coronary artery bypass grafting
Target vessel non-target lesion revascularisation | Baseline, 3 months, 6 months, 12 months
  Any lesion or revascularisation of a lesion in the target vessel other than the target lesion, respectively
Non-target vessel revascularisation | Baseline, 3 months, 6 months, 12 months
  Revascularisation of a vessel for which revascularisation is not attempted in the first place, or of one with no lesion with high-risk plaque characteristics.
Improvement in angina class as defined by the Canadian Cardiovascular Society (CCS) | Baseline, 3 months, 6 months, 12 months
  Any improvement in the angina class of the Canadian Cardiovascular Society (CCS) from a higher class to a lower class

OTHER OUTCOMES:
Procedural success | At the end of percutaneous coronary intervention procedure
  Achievement of < 30 % residual diameter stenosis of the target lesion assessed by visual inspection or QCA and no in-hospital major adverse cardiac events (MACE, a composite of death, MI, or repeat coronary revascularisation of the target lesion).

CONTACTS AND LOCATIONS:
Overall Officials: Barış İKİTİMUR, Study Director — İstanbul University-Cerrahpaşa, Cerrahpaşa School of Medicine
Locations (1):
- Istanbul University-Cerrahpaşa, Cerrahpaşa Faculty of Medicine, Prof. Dr. Murat Dilmener Hospital, Istanbul, Bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial
Supporting Information: Study Protocol, ICF
Time Frame: Starting from the publication of results and earning of the 1 year of publication